CLINICAL TRIAL: NCT04031391
Title: Effects of a Physical Exercise Program on Patients Affected With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7Z17/032
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Fibromyalgia
Keywords: physical activity; fibromyalgia; pain; exercice; quality of live
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized, multi-center, clinical trial composed of two groups response variables and a twelve weeks follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical activity group (Experimental)
  Interventions: Other: Physical activity
- Control group (No Intervention)

INTERVENTIONS:
Other: Physical activity — The intervention group: engaged in a therapeutic physical activity program involving low-intensity exercise, strength and balance work for 2 days a week over a 12-week period, with each session lasting 90 minutes. Both the intervention group and the control group separately completed the various baseline surveys which were part of the study. Once the intervention was over, they answered them again, also separately.
  The classes were led by an experienced physiotherapist who followed the physical exercise guidelines established by the American College of Sports Medicine (ACSM), although the intensity of the exercises was adapted to the participants' tolerance levels
  Arms: physical activity group

SUMMARY:
Physical activity has been used for a number of years in the treatment of fibromyalgia (FM). The main objective of this study is to compare the effects of physical activity on two groups of women diagnosed with fibromyalgia (FM) in terms of pain, quality of life and the impact of the condition on their daily lives. Methods: this was a randomized clinical trial to assess the effects of physical activity performed by subjects assigned to one of two groups on the scores of three questionnaires (the pain Visual Analogue Scale, the FIQ questionnaire and the SF-36 health questionnaire) administered before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Women

* Ages of 40 and 75
* Diagnosis fibromyalgia (code M79.7)
* Anoia region

Exclusion Criteria:

* Pregnant
* Unable to participate in the physical activity program.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
The visual analogue scale (VAS) | two months
  evaluate pain, with a score of 0 to 10
The Spanish version of the SF-36 questionnaire | two months
  used to assess their perceived state of health. It includes eight variables: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health
the Fibromyalgia Impact Questionnaire (FIQ) | two months
  measures physical functioning, ability to undertake work and general well-being, with a score from 0 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: JACOBO MENDIOROZ PEÑA, MD, Study Chair — Institut Catala de Salut
Locations (1):
- Espai Civic Centre, Igualada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No